CLINICAL TRIAL: NCT04355130
Title: Autologous Tansfusion REquirements in Bone MArrow Harvest: The ATREMA Study
Acronym: ATREMA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2916
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-03

CONDITIONS: Bone Marrow Donors
MeSH Terms: interventions — Iron; Vitamin B 12

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Iron, vitamin B12 and acid folic supplementation — Vitamin and iron supplementation is administered one-two weeks before donation, and consist of iron supplementation (i.v. infusion of 20 mg/Kg ferric carboxymaltose in saline 100 ml), s.c. injection of 1 mg of vitamin B12 and acid folic 5 mg/die per os until day +15 post BM donation. BM collection is carried out by the transplant team and a maximal dose of 20-22 ml/Kg of the donor body weight is collected under general anesthesia (induction with fentanyl 1-3 mcg/Kg, Propofol 2-3 mg/Kg, rocuronium 0,6 mg/Kg and mantenaince with sevoflurane 0,8 MAC). Noninvasive cardiac output, blood pressure and hemoglobin monitoring are carried out during the entire procedure and in in the recovery room using the ClearSight™ system (Edwards Clinical) and the Radical Pulse co oxymeter (Masimo). After discharge from the hospital, donors will be revaluated on day + 7 after BM collection, and blood tests will be repeated in outpatient setting.

SUMMARY:
Despite perioperative autologous donation (PAD) is widely used in healthy bone marrow (BM) donors to restrain the hemoglobin decrease after BM harvest, this practice is not supported by strong clinical evidences and has been abandoned by some transplant teams. The critical revision of data relative to 102 BM collection procedures performed at our center between 2014 and 2018 failed to demonstrate an advantage of 1 over 2 PAD. Conversely, clearly emerged that PAD reduce the hemoglobin levels at BM harvest. Basically, PAD practice consists in the transfer of RBCs from the subject into a plastic bag and back to the subject at BM harvesting. Indeed, the evidence of clinical benefits of PAD in BM donors are still elusive. For this reason, current procedures on unrelated donors recommend iron and vitamin supplementation before the BM harvest, but let the decision to perform or not PAD at collection centers. Detailed data on the safety and feasibility of BM harvest procedures in absence of PAD have been rarely reported. The investigators collect data on BM harvest in healthy donors who don't have PAD collected. The investigators expect that no allogeneic transfusions are required and that Hb levels after collection are similar to those recorded in the historical cohort gathered at the same center receiving 1 or 2 PAD.

ELIGIBILITY:
Inclusion Criteria:

* Familial donors qualified to donate BM hematopoietic stem cells and accepting to participate to this study

Exclusion Criteria:

* Any planned deviation connected with abnormalities in the health status and/or laboratory tests of the donor, even though it does not prevent him from donation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To collect data on BM harvest in healthy donors who don't have PAD collected. We expect that no allogeneic transfusions are required and that Hb levels after collection are similar to those recorded in our historical cohort receiving 1 or 2 PAD.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Hb values | during procedure
  Hb values recorded in healthy BM donors receiving iron and vitamins supplementation at the end of BM harvest

SECONDARY OUTCOMES:
Hb values | day 1 post BM harvest
  Hb values recorded in healthy BM donors receiving iron and vitamins supplementation at day 1 after BM harvest
Hb values | day 7 post BM harvest
  Hb values recorded in healthy BM donors receiving iron and vitamins supplementation at day 7 after BM harvest

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Teofili, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy